CLINICAL TRIAL: NCT06686186
Title: A Prospective Cohort of Hainan Community Elderly Population with Cognitive Impairment
Brief Title: Hainan Community Cognition Cohort
Status: Recruiting | Type: Observational
Sponsor: Hainan Medical College (Other)
Collaborators: The Second Affiliated Hospital of Hainan Medical University (Other); Xuanwu Hospital, Beijing (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Jindong Ding Petersen, Professor, Hainan Medical College
Other Study IDs: Hainan Medical University; ZDYF2024SHFZ064 (Other Grant/Funding Number: Hainan Provincial Department Of Science and Technology); 82360673 (Other Grant/Funding Number: National Natural Science Foundation of China); XRC2022005 (Other Grant/Funding Number: Hainan Medical University)
Record Dates: First submitted 2024-10-23; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Impairment; Dementia; Age Problems
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Plan to collect blood samples from some participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — There were no interventions in our cohort. The subjects of our cohort were and will be followed up at the regular intervals.

SUMMARY:
This is a community-based prospective cohort study in Hainan Province, China. The study was initialized in 2023 and included older residents for longitudinal follow-up. The research aims to identify risk factors as well as health and social outcomes that are associated with cognitive impairment in elderly populations, and independently develop AI-assisted software and applications for cognitive enhancement and physical rehabilitation training.

DETAILED DESCRIPTION:
This is a community-based prospective cohort study in Hainan Province, China. Subjects are individuals aged 60 years and above who have lived in the communities for more than six months and have signed informed consent. The research have been initialed in 2023 and aims to identify the risk factors associated with cognitive impairment, to develop software for cognitive enhancement and physical rehabilitation training. The study includes three steps: first, to conduct cognitive function screening in 16 communities in four districts (Xiuying, Meilan, Longhua, and Qiongshan) of Haikou City and establish a database for the elderly in tropical regions; second, to identify risk factors associated with cognitive impairment in the elderly population; finally, to independently develop a software for cognitive function enhancement and physical rehabilitation training.

ELIGIBILITY:
* Inclusion Criteria:

  * Age 60 years and above
  * Lived in the community for more than 6 months
  * Signed the informed consent form
* Exclusion Criteria:

  * Cannot complete the survey

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community residents aged 60 years or older in Hainan Province, China
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2053-12-31 (Estimated); Study Completion 2053-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence and incidence of cognitive impairment base on the communities | An average of 1 to 2 years
  Mild cognitive impairment was measured using a Chinese version Mini-Mental State Examination, which was collected by questionnaire. The minimum value of the Mini-Mental State Examination is 0, and the maximum value is 30, the higher the score, the better the cognition outcome.
The prevalence and incidence of dementia using a population-based survey | An average of 1 to 2 years
  Dementia was determined by diagnosis of hospitalization or Clinical Dementia Rating Scale (Montreal Cognitive Assessment, MoCA). The minimum value of the MoCA is 0, and the maximum value is 30, the higher the score, the better the outcome.
  In addition, subtypes of dementia will be based on the specific clinical diagnosis.
The conversion rate of normal to cognitive impairment | An average of 1 to 2 years
  Percentage of enrolled population that convert from normal to cognitive impairment
The conversion rate of cognitive impairment to dementia | An average of 1 to 2 years
  Percentage of enrolled population that convert from cognitive impairment to dementia

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan Medical University, Haikou, Hainan, China